CLINICAL TRIAL: NCT02595463
Title: Intravenous Lidocaine to Decrease Postoperative Pain in Pediatric Patients Undergoing Tonsillectomy: A Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Intravenous Lidocaine for Post-Tonsillectomy Pain in Pediatric Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Hubert Benzon, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-741
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): Following intraoperative IV placement, a 1.5 mg/kg bolus does of lidocaine hydrochloride is given and is followed by a continuous infusion of 2 mg/kg/hr until discharge from the Phase 1 recovery period.
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Following intraoperative IV placement, a bolus of saline is given and is followed by a continuous infusion until discharge from the Phase 1 recovery period. The volume of the bolus and rate of infusion are equivalent to that which would have been given in the experimental arm.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — Intraoperative dose of intravenous lidocaine followed by an infusion until discharge from the initial recovery period.
  Other Names: Xylocaine, Lidocaine Hydrochloride
  Arms: Lidocaine
Drug: Saline — Intraoperative dose of saline followed by an infusion until discharge from the initial recovery period.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether giving lidocaine intravenously during and after a tonsillectomy surgery is effective in decreasing postoperative pain.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether giving lidocaine intravenously during and after a tonsillectomy surgery is effective in decreasing postoperative pain when compared to placebo.

Participants will be in one of two arms. Those in Arm 1 will receive a lidocaine bolus and infusion throughout the initial recovery period while those in Arm 2 will receive an equal volume of normal saline. Subjects will be monitored and assessed for pain during their time in the hospital and followed up on at home for a week after the surgery. Primary outcomes will be measure of pain. Secondary outcome measures will include pain medication use, emergence delirium, incidence of laryngospasm, and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for Tonsillectomy (with or without Adenoidectomy) with Dr. Kathleen Billings or Dr. Stephen Hoff at Lurie Children's Hospital
* American Society of Anesthesiology (ASA) patient classification I-III (Healthy patient to a patient with mild systemic disease)

Exclusion Criteria:

* Physical or developmental delays
* Psychiatric illness
* Current use of sedative or anticonvulsant medications
* Pre-existing renal disease (ranging from stage 2 [mild] to stage 5 [end stage])
* Pre-existing cardiovascular disease (including, not limited to congenital heart disease or arrythmia)
* Pre-existing liver disease
* Pre-existing cerebral or neuromuscular disease
* Patient or family history of Malignant Hyperthermia
* Recent history of upper respiratory infection within last 7 days
* Regular use of analgesic medication
* Diagnosis of severe obstructive sleep apnea requiring overnight stay for observation
* Other procedure scheduled in addition to tonsillectomy
* History of allergies to local anesthetics

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2015-11; Primary Completion 2024-06-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Observer Rated Pain Intensity | Within the immediate post-operative period (90 minutes after surgery)
  Observer Rated Pain Intensity will be measured using the Children's Eastern Ontario Pain Scale (CHEOPS) at regular 5 and 15 minute time intervals.

SECONDARY OUTCOMES:
Patient Rated Pain Intensity | Within the immediate post-operative period (90 minutes after surgery)
  Patient Rated Pain Intensity will be measured using the Faces Pain Scale - Revised (FPS-R) by pointing to pictures of faces displaying a spectrum of pain at regular 5 and 15 minute time intervals.
Observer Rated Emergence Delirium | Within the immediate post-operative period (90 minutes after surgery)
  Observer Rated Emergence Delirium will be measured using the he Pediatric Emergence Delirium (PAED) Scale at regular 5 and 15 minute time intervals.
Observer Rated PACU Discharge Criteria | Within the immediate post-operative period (90 minutes after surgery)
  Observer Rated PACU Discharge Criteria will be measured using the modified Aldrete Scale at regular time intervals.
Parent Rated Postoperative Pain at Home | Every day, up to 7 days postoperatively
  Parent Rated Postoperative Pain at Home will be measured using the Parents Postoperative Pain Measures (PPPM) questionnaire and Numerical Rating Scale to report on the intensity of their child's pain.
Medication Journal | Every day, up to 7 days postoperatively
  Parents will keep a journal of all pain medication given to their children to treat pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Benzon, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Weibel S. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Database Syst Rev. 2015 Jul 16;(7):CD009642. doi: 10.1002/14651858.CD009642.pub2. PMID 26184397
- [Background] Koppert W, Ostermeier N, Sittl R, Weidner C, Schmelz M. Low-dose lidocaine reduces secondary hyperalgesia by a central mode of action. Pain. 2000 Mar;85(1-2):217-24. doi: 10.1016/s0304-3959(99)00268-7. PMID 10692621
- [Background] Goldman JL, Baugh RF, Davies L, Skinner ML, Stachler RJ, Brereton J, Eisenberg LD, Roberson DW, Brenner MJ. Mortality and major morbidity after tonsillectomy: etiologic factors and strategies for prevention. Laryngoscope. 2013 Oct;123(10):2544-53. doi: 10.1002/lary.23926. Epub 2013 Apr 17. PMID 23595509
- [Background] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581